CLINICAL TRIAL: NCT05213286
Title: The Development of a Screening Questionnaire to Discriminate Autism Spectrum Disorder and Schizotypal Disorder, and Validation of the Danish Version of RAADS-R
Acronym: ZA-RAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Rizwan Parvaiz, Medical doctor, Director of Autism Research, Glostrup University Hospital, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZA-RAA
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Autism Spectrum Disorder; Schizotypal Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Schizotypal Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients referred for assessment of ASD, non-ASD psychiatric patients and control group (Other): All three groups will be tested with RAADS-R-DK and ZAQ. The results from these diagnostic tests will be compared to gold standard clinical assessments in specialized multidisciplinary teams
  Interventions: Diagnostic Test: Application of ZAQ and RAADS-R-DK

INTERVENTIONS:
Diagnostic Test: Application of ZAQ and RAADS-R-DK — Test of the questionnaires in each of the three groups.

SUMMARY:
The aim of the study is to investigate the validity, reliability and clinical features of a Danish version of the Ritvo Autism Asperger Diagnostic Scale-Revised (RAADS-R). A self-reporting scale devise used as a supplementary questionnaire in diagnosing autism spectrum disorder (ASD) in adults. Furthermore the validity of novel screening questionnaire: SchiZotypal Autism Questionnaire (ZAQ), will be investigated. ZAQ is developed to discriminate Schizotypal Disorder from ASD.

DETAILED DESCRIPTION:
The study has 2 parts.

Part 1:

The objective is to develop and validate a self-report screening questionnaire to efficiently discriminate between Schizotypal Disorder (SD) and Autism Spectrum Disorder (ASD) within the adult population. Discriminating ASD from SD in a clinical setting is a complex and time-consuming task, as they share considerable features both at the symptomatic and the diagnostic criteria. A pilot version of this questionnaire have been developed with 139 questions and named schiZotypy Autism Questionnaire (ZAQ), to discriminate between these conditions.

Part 2:

RAADS-R scale, which is a clinical tool that aims to better identify autism spectrum disorders The scale is a self-administered questionnaire completed by the patient himself assisted by a clinician (psychiatrist, psychologist) which ensures the understanding of issues and the choice of answers. The scale contains 80 items including 64 questions describe specific symptoms of autism spectrum disorders and 16 questions to describe non-symptomatic behaviors.

The objective of this study is to perform a complete validation of this scale in a Danish translation.

For both parts of the study 600 adults will be included, 200 adults referred for assessment of autism, 200 adults with another psychiatric disorder, and 200 adults without psychiatric disease.

ELIGIBILITY:
Inclusion Criteria:

1. Al patient referred to the outpatient clinic for ADHD and Autism at PCG, in the research period, for diagnostic assessment of Autism Spectrum Disorder (Pervasive Developmental Disorder, infantile autism, atypical autism and Asperger Syndrome)
2. WAIS > 85, or Raven or no-clinical suspicion and education level of 11 years or above
3. Completion of

   1. Clinical assessment
   2. Adult Asperger Assessment (AAA)
   3. Psychopathology evaluation using DSM-V
   4. A conclusion based on interdisciplinary consensus

Exclusion Criteria:

1. Insufficient Danish language skills
2. Acute psychiatric illness prompting departure/dismissal from the diagnostic assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
ZAQ | up to 1 month
  schiZotypy Autism Questionnaire
RAADS-R-DK | Up to 1 month
  Ritvo Autism Asperger Diagnostic Scale-Revised-Danish version

SECONDARY OUTCOMES:
AQ | Up to 1 month
  Autism Quotient
WHO-DAS 2.0 | Up to 1 month
  Assessment instrument for health and disability.
WHO-5 | Up to 1 month
  Assessment of psychological well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Glostrup University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parvaiz R, Vindbjerg E, Crespi B, Happe F, Schalbroeck R, Al-Sayegh Z, Danielsen IM, Tonge B, Videbech P, Abu-Akel A. Protocol for the development and testing of the schiZotypy Autism Questionnaire (ZAQ) in adults: a new screening tool to discriminate autism spectrum disorder from schizotypal disorder. BMC Psychiatry. 2023 Mar 28;23(1):200. doi: 10.1186/s12888-023-04690-3. PMID 36978026
- [Derived] Parvaiz R, Al-Sayegh Z, Jacobsen PK, Danielsen IM, Videbech P. Validation of a screening tool for autism spectrum disorder in adults - a study protocol. Dan Med J. 2022 Nov 23;69(12):A02220118. PMID 36458608